CLINICAL TRIAL: NCT03620448
Title: Immediate Treatment Outcomes of Bubble-cpap Versus Oxygen Therapy in Preterm Babies Presenting With Respiratory Distress Syndrome at Kilimanjaro Christian Medical Center
Brief Title: Immediate Treatment Outcomes of b-CPAP vs Oxygen Therapy in Preterm Babies Presenting With RDS at KCMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kilimanjaro Christian Medical Centre, Tanzania (Other)
Responsible Party: Principal Investigator, Dr. Annette M Baine, Principal Investigator, Kilimanjaro Christian Medical Centre, Tanzania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPAP1
Record Dates: First submitted 2018-07-02; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Respiratory Distress Syndrome in Premature Infant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- bCPAP Arm. (Experimental): Babies randomized to receive bCPAP were started (by principle investigator assisted by a clinician) on bCPAP (Rice 360◦c low cost bCPAP device) consisting of 3 components:
  (i) An oxygen concentrator with a gas flow fate of 3-4L/min, (ii) A nasal interface (short nasal prongs) connecting the baby's airway to a two limb circuit i.e the inspiratory limb connected to the bCPAP machine and the expiratory limb connected to the water bottle and (iii) An expiratory limb with the distal end submerged 6cm in water to generate an end expiratory pressure as seen in appendix 7. adopted from suppliers of the pumani bCPAP machine in Kenya.
  Interventions: Device: bCPAP Arm
- Oxygen Arm (Other): Preterms on the control arm and those whose parents didn't consent received the standard treatment for RDS i.e pure oxygen via nasal prongs from the oxygen cylinders.
  Interventions: Other: Oxygen Arm

INTERVENTIONS:
Device: bCPAP Arm — bCPAP (Rice 360◦c low cost bCPAP device)
  Arms: bCPAP Arm.
Other: Oxygen Arm — Oxygen therapy from oxygen cylinders
  Arms: Oxygen Arm

SUMMARY:
Bubble - Continuous positive airway pressure (CPAP) has been reported to be effective, cheaper, simpler and more accessible compared to mechanical ventilator and surfactant treatment for preterms with respiratory distress syndrome in the neighbouring countries. This study aims to implement and determine the effectiveness of bCPAP and its immediate outcomes compared to oxygen therapy in preterm babies presenting with respiratory distress syndrome (RDS).

DETAILED DESCRIPTION:
Effective treatment of preterm babies with RDS requires exogenous surfactant and/or mechanical ventilation but these are of limited availability in developing countries.

bCPAP is generated by exhalation against a constant opening pressure that produces positive end-expiratory pressure. This in-turn helps in maintaining lung volume at the end of expiration, preventing atelectasis, improving oxygenation, reducing respiratory fatigue and eventually preventing respiratory failure. bCPAP (Rice 360◦c low cost bCPAP device) consisting of 3 components: : (i)An air compressor connected to an oxygen concentrator with a gas flow fate of 3-4 L/min; (ii) A nasal interface (short nasal prongs) connecting the baby's airway to a two limb circuit i.e the inspiratory limb connected to the bCPAP machine and the expiratory limb connected to the water bottle and; (iii) An expiratory limb with the distal end submerged 6 cm in water to generate an end expiratory pressure

At the neonatal unit at Kilimanjaro Christian Medical Center (KCMC), the standard of care for Preterm babies with RDS is receiving oxygen therapy via nasal prongs from oxygen cylinders.

ELIGIBILITY:
Inclusion Criteria:

* All preterm babies (< 37 weeks of gestation determined using Finnstorm score) presenting with signs of RDS (tachypnea of >60breaths /min, intercostal and subcostal recessions, nasal flaring, grunting and cyanosis)

Exclusion Criteria:

* Preterm babies with birthweight less than 1kg (bCPAP machine can only be used in babies with body weight of 1-10kg)
* Congenital malformations (cleft palate and lip, tracheal esophageal fistula and diaphragmatic hernia)
* Mothers who refused to consent

Ages: 28 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Comparing the number of babies that survived with bCPAP treatment versus Oxygen therapy | 6 months
  The proportion of babies discharged alive in the bCPAP arm versus the oxygen therapy arm.

SECONDARY OUTCOMES:
Treatment duration | 6 months
  The time spent on the allocated treatment arm till RDS symptoms (tachypnea (>60breaths/min), intercostal and subcostal recessions, nasal flaring, grunting and cyanosis) resolve.
Duration of hospital stay | 6 months
  Time from admission into the neonatal ward to discharge (dead or alive).
Treatment complications | 6 months
  Whilst the subject is receiving treatment, the following complications will be observed and recorded; like pneumothorax, nasal bleeding, injury to the skin, nose or eye, aspiration pneumonia, vomiting and any other complication considered related to the treatment as per the principal investigator's clinical judgement.

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be shared as per the local country guidelines.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be made available 12 months after study completion.
Access Criteria: Persons requesting data will be asked to sign a data transfer agreement as well as provide evidence of ethical clearance.

REFERENCES:
- [Result] Kawaza K, Machen HE, Brown J, Mwanza Z, Iniguez S, Gest A, Smith EO, Oden M, Richards-Kortum RR, Molyneux E. Efficacy of a low-cost bubble CPAP system in treatment of respiratory distress in a neonatal ward in Malawi. PLoS One. 2014 Jan 29;9(1):e86327. doi: 10.1371/journal.pone.0086327. eCollection 2014. PMID 24489715